CLINICAL TRIAL: NCT02114697
Title: Accelerated Atherosclerosis in High Risk Population Groups: An Assessment by Magnetic Resonance Imaging
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped when the original principal investigator moved to a new institution.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, John Oshinski, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00059784
Record Dates: First submitted 2014-04-10; First posted 2014-04-15 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Atherosclerosis
Keywords: Cancer survivorship; Cardiovascular disease; Stroke; Transient ischemic attack (TIA)
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Stroke; Ischemic Attack, Transient | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: The protocol originally specified randomizing participants to a study arm, but the protocol was amended to clarify that a participant's cardiologist could change the treatment regimens that participants were assigned to so that no participant was restricted from statin therapy.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lifestyle modification (Active Comparator): Lifestyle modification is tailored to each participant and includes a recommended exercise regimen, a healthy diet and decreasing alcohol intake.
  Interventions: Behavioral: Lifestyle modification
- Statin therapy (Experimental): Participants will receive statin medication along with instruction about regular exercise.
  Interventions: Drug: Statin therapy

INTERVENTIONS:
Drug: Statin therapy — Statin therapy includes rosuvastatin 20 mg administered orally, once a day, for the duration of the trial, which is 3 years. Participants may also receive a different type of statin as prescribed by their cardiologist based on clinical judgement.
  Other Names: Crestor
  Arms: Statin therapy
Behavioral: Lifestyle modification — Lifestyle modification includes a recommended exercise regimen, a healthy diet and decreasing alcohol intake for 3 years.
  Arms: Lifestyle modification

SUMMARY:
The goal of this study is to assess a slimy substance that settles/deposits along blood vessel wall. This slimy substance is called plaque. Plaque could be made up of fat, calcium or both. Plaque deposition narrows the vessels. This leads to decreased blood flow to various parts of body. Blood vessels include vessels that supply to heart (coronary), vessels to brain (carotid), vessels to kidneys (renal) and vessels to legs (femoral). Decreased blood flow causes symptoms such as brain stroke, heart attack, leg pain. Similarly individuals at risk of cardiovascular disease can have certain markers elevated in their blood that can be measured by simple blood tests.

High or increased plaque deposition is seen in neck vessels of cancer patients who received radiation to chest or head and neck as part of their cancer treatment. Cancer survivors are at increased risk of plaque development and are therefore called high-risk population. Exercise +/- fat lowering medicine can potentially decrease plaque deposition and statins are one of the several fat lowering medications.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) and cancer are the leading causes of suffering and death amongst the American population. While an ever-increasing number of cancer survivors have a favorable outcome due to advances in cancer treatment; cancer survivors remain at high risk of developing CVD at an early age. There is scant information available on the pathogenic process that contributes to cardiovascular threat amongst cancer survivors and little is known about the interventions, which may interrupt or decrease the risk of CVD in this population. Importantly, early-subclinical markers may substantially precede clinical markers.

The objective of this project is to accurately determine the constituents and characteristics of atherosclerotic plaques in carotid arteries by magnetic resonance imaging (MRI) techniques in cancer survivors; at different data intervals: before and after administration of treatment (medical and life style modification) and then correlate contrast agent dynamics with serum markers of inflammation and other tests of cardiac or vascular dysfunction, where available.

The proposed study involves 100 asymptomatic patients who received prior chest or head and neck radiation therapy (HNXRT) as part of cancer treatment. MRI data (direct assessment of atherosclerosis) would be correlated with indirect measures of atherosclerosis (blood surrogate markers & metabolomics).

The investigators intend to conduct an initial baseline MRI, blood tests (to correlate with surrogate markers of inflammation) and other tests whenever available of cardiac or vascular dysfunction. This cohort will be followed up with medication and/or life style modification regimen for a period of initially18 months and subsequently at 36 months. A repeat of all baseline studies (MRI and blood tests) would be performed as part of the 18 and 36-month follow-up. The plaque characteristics found at MRI will be correlated with results of blood tests (baseline, 18 and 36 months) and changes in one or both will be the expected end point of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 22 and above with prior head and neck or chest irradiation
* Six months or more post head and neck irradiation
* Documented subclinical cardiovascular disease (inflammatory markers in the serum)
* Pre-existing plaques (detected by ultrasound, CT or MRI)
* Asymptomatic major arterial stenosis
* Not being considered for arterial surgery or endovascular treatment.

Exclusion Criteria:

* Recurrence of cancer (with or without treatment)
* Planned surgical or endovascular intervention for revascularization of carotid arteries at the time of enrollment
* Renal failure
* Estimated glomerular filtration rate (eGFR) < 45 (calculation based on serum creatinine levels, race, age and gender)
* Medically unstable or hematologic, renal, or hepatic dysfunction
* Non-atherosclerotic arterial stenosis (dissection)
* Presence of stents or external clips that can cause artifacts impairing accurate interpretation of MRI data
* Contraindications to MRI: cardiac pacemaker, metal implants, metal in eyes, pregnant or nursing women, claustrophobia, allergy to MRI contrast
* Physical or mental impairment that would limit the patient's ability to comply with the medical instructions or study procedures

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-04; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Oshinski, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Background] Ota H, Yu W, Underhill HR, Oikawa M, Dong L, Zhao X, Polissar NL, Neradilek B, Gao T, Zhang Z, Yan Z, Guo M, Zhang Z, Hatsukami TS, Yuan C. Hemorrhage and large lipid-rich necrotic cores are independently associated with thin or ruptured fibrous caps: an in vivo 3T MRI study. Arterioscler Thromb Vasc Biol. 2009 Oct;29(10):1696-701. doi: 10.1161/ATVBAHA.109.192179. Epub 2009 Jul 16. PMID 19608971
- [Background] Virmani R, Burke AP, Kolodgie FD, Farb A. Vulnerable plaque: the pathology of unstable coronary lesions. J Interv Cardiol. 2002 Dec;15(6):439-46. doi: 10.1111/j.1540-8183.2002.tb01087.x. PMID 12476646
- [Background] Yeh JM, Nekhlyudov L, Goldie SJ, Mertens AC, Diller L. A model-based estimate of cumulative excess mortality in survivors of childhood cancer. Ann Intern Med. 2010 Apr 6;152(7):409-17, W131-8. doi: 10.7326/0003-4819-152-7-201004060-00005. PMID 20368646
- [Background] Dorresteijn LD, Kappelle AC, Boogerd W, Klokman WJ, Balm AJ, Keus RB, van Leeuwen FE, Bartelink H. Increased risk of ischemic stroke after radiotherapy on the neck in patients younger than 60 years. J Clin Oncol. 2002 Jan 1;20(1):282-8. doi: 10.1200/JCO.2002.20.1.282. PMID 11773180
- [Background] Jordan LC, Duffner PK. Early-onset stroke and cerebrovascular disease in adult survivors of childhood cancer. Neurology. 2009 Dec 1;73(22):1816-7. doi: 10.1212/WNL.0b013e3181c33b10. Epub 2009 Oct 21. No abstract available. PMID 19846829
- [Background] Diller L, Chow EJ, Gurney JG, Hudson MM, Kadin-Lottick NS, Kawashima TI, Leisenring WM, Meacham LR, Mertens AC, Mulrooney DA, Oeffinger KC, Packer RJ, Robison LL, Sklar CA. Chronic disease in the Childhood Cancer Survivor Study cohort: a review of published findings. J Clin Oncol. 2009 May 10;27(14):2339-55. doi: 10.1200/JCO.2008.21.1953. Epub 2009 Apr 13. No abstract available. PMID 19364955
- [Background] Mertens AC, Yasui Y, Neglia JP, Potter JD, Nesbit ME Jr, Ruccione K, Smithson WA, Robison LL. Late mortality experience in five-year survivors of childhood and adolescent cancer: the Childhood Cancer Survivor Study. J Clin Oncol. 2001 Jul 1;19(13):3163-72. doi: 10.1200/JCO.2001.19.13.3163. PMID 11432882
- [Background] Haynes JC, Machtay M, Weber RS, Weinstein GS, Chalian AA, Rosenthal DI. Relative risk of stroke in head and neck carcinoma patients treated with external cervical irradiation. Laryngoscope. 2002 Oct;112(10):1883-7. doi: 10.1097/00005537-200210000-00034. PMID 12368635
- [Background] Bowers DC, Liu Y, Leisenring W, McNeil E, Stovall M, Gurney JG, Robison LL, Packer RJ, Oeffinger KC. Late-occurring stroke among long-term survivors of childhood leukemia and brain tumors: a report from the Childhood Cancer Survivor Study. J Clin Oncol. 2006 Nov 20;24(33):5277-82. doi: 10.1200/JCO.2006.07.2884. Epub 2006 Nov 6. PMID 17088567
- [Background] Moser EC, Noordijk EM, van Leeuwen FE, le Cessie S, Baars JW, Thomas J, Carde P, Meerwaldt JH, van Glabbeke M, Kluin-Nelemans HC. Long-term risk of cardiovascular disease after treatment for aggressive non-Hodgkin lymphoma. Blood. 2006 Apr 1;107(7):2912-9. doi: 10.1182/blood-2005-08-3392. Epub 2005 Dec 8. PMID 16339404
- [Background] Steele SR, Martin MJ, Mullenix PS, Crawford JV, Cuadrado DS, Andersen CA. Focused high-risk population screening for carotid arterial stenosis after radiation therapy for head and neck cancer. Am J Surg. 2004 May;187(5):594-8. doi: 10.1016/j.amjsurg.2004.01.014. PMID 15135672
- [Background] Casscells W, Naghavi M, Willerson JT. Vulnerable atherosclerotic plaque: a multifocal disease. Circulation. 2003 Apr 29;107(16):2072-5. doi: 10.1161/01.CIR.0000069329.70061.68. No abstract available. PMID 12719287
- [Background] Hatsukami TS, Ross R, Polissar NL, Yuan C. Visualization of fibrous cap thickness and rupture in human atherosclerotic carotid plaque in vivo with high-resolution magnetic resonance imaging. Circulation. 2000 Aug 29;102(9):959-64. doi: 10.1161/01.cir.102.9.959. PMID 10961958
- [Background] MacNeill BD, Lowe HC, Takano M, Fuster V, Jang IK. Intravascular modalities for detection of vulnerable plaque: current status. Arterioscler Thromb Vasc Biol. 2003 Aug 1;23(8):1333-42. doi: 10.1161/01.ATV.0000080948.08888.BF. Epub 2003 Jun 12. PMID 12805071
- [Background] Crisby M, Nordin-Fredriksson G, Shah PK, Yano J, Zhu J, Nilsson J. Pravastatin treatment increases collagen content and decreases lipid content, inflammation, metalloproteinases, and cell death in human carotid plaques: implications for plaque stabilization. Circulation. 2001 Feb 20;103(7):926-33. doi: 10.1161/01.cir.103.7.926. PMID 11181465
- [Background] Davies MJ. Stability and instability: two faces of coronary atherosclerosis. The Paul Dudley White Lecture 1995. Circulation. 1996 Oct 15;94(8):2013-20. doi: 10.1161/01.cir.94.8.2013. No abstract available. PMID 8873680
- [Background] Kolodgie FD, Virmani R, Burke AP, Farb A, Weber DK, Kutys R, Finn AV, Gold HK. Pathologic assessment of the vulnerable human coronary plaque. Heart. 2004 Dec;90(12):1385-91. doi: 10.1136/hrt.2004.041798. No abstract available. PMID 15547008
- [Background] Hansson GK. Inflammation, atherosclerosis, and coronary artery disease. N Engl J Med. 2005 Apr 21;352(16):1685-95. doi: 10.1056/NEJMra043430. No abstract available. PMID 15843671
- [Background] Krams R, Segers D, Mousavi Gourabi B, Maat W, Cheng C, van Pelt C, van Damme LC, de Feyter P, van der Steen T, de Korte CL, Serruys PW. Inflammation and atherosclerosis: mechanisms underlying vulnerable plaque. J Interv Cardiol. 2003 Apr;16(2):107-13. doi: 10.1046/j.1540-8183.2003.08021.x. No abstract available. PMID 12768913
- [Background] Libby P. Inflammation in atherosclerosis. Nature. 2002 Dec 19-26;420(6917):868-74. doi: 10.1038/nature01323. PMID 12490960
- [Background] Hansson GK, Robertson AK, Soderberg-Naucler C. Inflammation and atherosclerosis. Annu Rev Pathol. 2006;1:297-329. doi: 10.1146/annurev.pathol.1.110304.100100. PMID 18039117
- [Background] Libby P, Ridker PM, Maseri A. Inflammation and atherosclerosis. Circulation. 2002 Mar 5;105(9):1135-43. doi: 10.1161/hc0902.104353. PMID 11877368
- [Background] Stone GW, Maehara A, Lansky AJ, de Bruyne B, Cristea E, Mintz GS, Mehran R, McPherson J, Farhat N, Marso SP, Parise H, Templin B, White R, Zhang Z, Serruys PW; PROSPECT Investigators. A prospective natural-history study of coronary atherosclerosis. N Engl J Med. 2011 Jan 20;364(3):226-35. doi: 10.1056/NEJMoa1002358. PMID 21247313
- [Background] Bengel FM. Vascular FDG uptake: further steps toward clinical acceptance. J Nucl Cardiol. 2008 Mar-Apr;15(2):154-6. doi: 10.1016/j.nuclcard.2008.01.010. No abstract available. PMID 18371583
- [Background] Croce K, Libby P. Intertwining of thrombosis and inflammation in atherosclerosis. Curr Opin Hematol. 2007 Jan;14(1):55-61. doi: 10.1097/00062752-200701000-00011. PMID 17133101
- [Background] Silvera SS, Aidi HE, Rudd JH, Mani V, Yang L, Farkouh M, Fuster V, Fayad ZA. Multimodality imaging of atherosclerotic plaque activity and composition using FDG-PET/CT and MRI in carotid and femoral arteries. Atherosclerosis. 2009 Nov;207(1):139-43. doi: 10.1016/j.atherosclerosis.2009.04.023. Epub 2009 Apr 24. PMID 19467659
- [Background] Fayad ZA, Fuster V. Characterization of atherosclerotic plaques by magnetic resonance imaging. Ann N Y Acad Sci. 2000 May;902:173-86. doi: 10.1111/j.1749-6632.2000.tb06312.x. PMID 10865837
- [Background] Mitsumori LM, Hatsukami TS, Ferguson MS, Kerwin WS, Cai J, Yuan C. In vivo accuracy of multisequence MR imaging for identifying unstable fibrous caps in advanced human carotid plaques. J Magn Reson Imaging. 2003 Apr;17(4):410-20. doi: 10.1002/jmri.10264. PMID 12655579
- [Background] Yuan C, Mitsumori LM, Beach KW, Maravilla KR. Carotid atherosclerotic plaque: noninvasive MR characterization and identification of vulnerable lesions. Radiology. 2001 Nov;221(2):285-99. doi: 10.1148/radiol.2212001612. PMID 11687667
- [Background] Ridker PM, Danielson E, Fonseca FA, Genest J, Gotto AM Jr, Kastelein JJ, Koenig W, Libby P, Lorenzatti AJ, MacFadyen JG, Nordestgaard BG, Shepherd J, Willerson JT, Glynn RJ; JUPITER Study Group. Rosuvastatin to prevent vascular events in men and women with elevated C-reactive protein. N Engl J Med. 2008 Nov 20;359(21):2195-207. doi: 10.1056/NEJMoa0807646. Epub 2008 Nov 9. PMID 18997196
- [Background] Courneya KS, Stevinson C, McNeely ML, Sellar CM, Friedenreich CM, Peddle-McIntyre CJ, Chua N, Reiman T. Effects of supervised exercise on motivational outcomes and longer-term behavior. Med Sci Sports Exerc. 2012 Mar;44(3):542-9. doi: 10.1249/MSS.0b013e3182301e06. PMID 21814149
- [Background] Ahmed HM, Blaha MJ, Nasir K, Rivera JJ, Blumenthal RS. Effects of physical activity on cardiovascular disease. Am J Cardiol. 2012 Jan 15;109(2):288-95. doi: 10.1016/j.amjcard.2011.08.042. Epub 2011 Oct 18. PMID 22011559
- [Background] Williams MA, Ades PA, Hamm LF, Keteyian SJ, LaFontaine TP, Roitman JL, Squires RW. Clinical evidence for a health benefit from cardiac rehabilitation: an update. Am Heart J. 2006 Nov;152(5):835-41. doi: 10.1016/j.ahj.2006.05.015. PMID 17070142
- [Background] Pannu N, Tonelli M. Strategies to reduce the risk of contrast nephropathy: an evidence-based approach. Curr Opin Nephrol Hypertens. 2006 May;15(3):285-90. doi: 10.1097/01.mnh.0000222696.92088.28. PMID 16609296

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 11 individuals gave informed consent to participate in the study, however, one withdrew from the study and one was lost to follow up before being assigned to a study arm. These individuals are not considered as enrolled as no clinical data were collected. Nine participants were assigned to a study arm and began the intervention.
Groups:
- Lifestyle Modification: Participants receiving information about lifestyle modifications including a recommended exercise regimen, a healthy diet and decreasing alcohol intake.
- Statin Therapy: Participants receiving statin therapy. A participant's cardiologist could change the treatment regimen that a participant was assigned to so that no participant was restricted from statin therapy. The results reflect the treatment each participant actually received rather than the treatment each participant was randomized to.
Period: Overall Study
Arm/Group | Lifestyle Modification | Statin Therapy
Started | 5 | 4
Completed Month 18 Visit | 0 | 1
Completed | 0 | 0
Not Completed | 5 | 4
Not completed — Study terminated | 5 | 4

BASELINE CHARACTERISTICS:
Population: All participants who began the intervention are included in the baseline analysis population description.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Modification | Statin Therapy | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.60 (3.64) | 62.25 (1.70) | 61.33 (2.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Plaque Volume of Carotid Arteries
Description: Plaque volume of carotid arteries were measured by MRI as a surrogate for progression of cardiovascular disease. Plaque volume varies with observed ranges from other studies ranging from 23.9 to 604.1mm^3. Plaque volume tends to increase with age. Increased plaque volume has an increased risk of vascular events.
Time Frame: Baseline, 18 months, 36 months
Population: This analysis includes all participants who completed the MRI at each time point. Most participants did not return for the follow up MRI measurements.
Measure: Mean (Standard Deviation); unit: Cubic millimeter (mm^3)
Arm/Group | Lifestyle Modification | Statin Therapy
Number analyzed (Participants) | 5 | 4
Cubic millimeter (mm^3)
  Baseline | 125.18 (8.09) | 108.88 (5.27)
  Month 18: number analyzed (Participants) | 0 | 1
  Month 18 |  | 114.70 (0.0)
  Month 36: number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the participant signed the consent form through the duration of participation (up to 36 months).
Description: All adverse events were graded as to their attribution (unrelated to protocol, or possibly, probably, or definitely related to protocol). All serious or unexpected adverse experiences and all deaths were recorded and reported according to the National Cancer Institute Common Toxicity Criteria. Serious adverse events were not expected to occur in this study due to the low risk involved with the study procedures performed.
Arm/Group | Lifestyle Modification | Statin Therapy
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT02114697/Prot_SAP_000.pdf